CLINICAL TRIAL: NCT00001567
Title: A Phase II Efficacy Study of Roferon-A in Hairy Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970060; 97-C-0060
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-04

CONDITIONS: Hairy Cell Leukemia
Keywords: Follow-Up Study; Relapse-Free Survival; Serum Soluble IL-2 Receptor; Hematologic Malignancy; Chronic Therapy
MeSH Terms: conditions — Leukemia, Hairy Cell; Hematologic Neoplasms | interventions — Interferon alpha-2

INTERVENTIONS:
Drug: Roferon-A

SUMMARY:
This study began as an efficacy study of interferon alpha-2a in patients with hairy cell leukemia. It was observed that most patients responded with interferon, but that very few complete responses were being obtained. Studies being done elsewhere confirmed the low complete remission rate. Once interferon was stopped, nearly uniformly disease progression requiring reinstitution of therapy was observed. There appear to be very few if any patients who will not require further therapy after receiving 12 or 18 months of continuous interferon treatment. Because of these findings, and in order to evaluate the safety and efficacy of long-term recombinant interferon-alpha (IFN-Alpha) in patients with hairy cell leukemia, we opted to administer interferon continuously to patients who were initially responsive to this drug. Of the 53 evaluable patients (of the 56 entered on this study), there was one complete remission, 41 partial remissions, 1 minor response, 9 patients with stable disease and only 1 patient with disease progression. Fourteen patients continue to receive interferon without interruption with a median duration of continuous interferon treatment of 9.2 years. Thirty-four patients discontinued interferon for a variety of reasons, the most common being the development of acquired interferon resistance in association with interferon antibodies. The resistance to interferon was manifested early, in the first 18 months of treatment, except in two cases. An important finding in this study is the continued slow, but significant, hematologic improvement in absolute granulocyte and platelet counts beyond 18 months of therapy, thereby indicating that prolonged treatment results in continued benefit rather than the production of antibodies with subsequent development of interferon resistance. Although it is clear from this study that hairy cell leukemia can be controlled in the long-term with interferon, longer follow-up will be necessary to determine if continuous therapy with interferon is better than intermittent therapy. The optimal therapy for hairy cell leukemia remains open to discussion. Although early reports suggested that 2-chlorodeoxyadenosine was curative, additional studies with longer periods of follow up suggests that as many as 30% of patients will relapse. This study provides the only instance where continuous long term treatment with interferon has been evaluated. This provides an opportunity to evaluate the long term toxicity of chronic interferon therapy, the long term efficacy of this treatment and to evaluate the potential benefits of long term interferon in preventing second malignancies, a complication noted in about 15% of patients treated in other fashions.

After their initial clinical evaluation, patients were given 3 million units of recombinant IFN-Alpha subcutaneously daily for 4 to 6 months. In responding patients, maintenance therapy was given at a dose of three million units subcutaneously 3 times per week. Responding patients have continued on therapy indefinitely.

DETAILED DESCRIPTION:
This study began as an efficacy study of interferon alpha-2a in patients with hairy cell leukemia. It was observed that most patients responded with interferon, but that very few complete responses were being obtained. Studies being done elsewhere confirmed the low complete remission rate. Once interferon was stopped, nearly uniform disease progression requiring reinstitution of therapy was observed. There appears to be very few if any patients who will not require further therapy after receiving 12 or 18 months of continuous interferon treatment. Because of these findings, and in order to evaluate the safety and efficacy of long-term recombinant interferon-alpha (IFN-Alpha) in patients with hairy cell leukemia, we opted to administer interferon continuously to patients who were initially responsive to this drug. Of the 53 evaluable patients (of the 56 entered on this study), there was one complete remission, 41 partial remissions, 1 minor response, 9 patients with stable disease and only 1 patient with disease progression. Fourteen patients continue to receive interferon without interruption with a median duration of continuous interferon treatment of 9.2 years. Thirty-four patients discontinued interferon for a variety of reasons, the most common being the development of acquired interferon resistance in association with interferon antibodies. The resistance to interferon was manifested early, in the first 18 months of treatment, except in two cases. An important finding in this study is the continued slow, but significant, hematologic improvement in absolute granulocyte and platelet counts beyond 18 months of therapy, thereby indicating that prolonged treatment results in continued benefit rather than the production of antibodies with subsequent development of interferon resistance. Although it is clear from this study that hairy cell leukemia can be controlled in the long-term with interferon, longer follow-up will be necessary to determine if continuous therapy with interferon is better than intermittent therapy. The optimal therapy for hairy cell leukemia remains open to discussion. Although early reports suggested that 2-chlorodeoxyadenosine was curative, additional studies with longer periods of follow up suggest that as many as 30% of patients will relapse. This study provides the only instance where continuous long term treatment with interferon has been evaluated. This provides an opportunity to evaluate the long term toxicity of chronic interferon therapy, the long term efficacy of this treatment and to evaluate the potential benefits of long term interferon in preventing second malignancies, a complication noted in about 15% of patients treated in other fashions.

After their initial clinical evaluation, patients were given 3 million units of recombinant IFN-Alpha subcutaneously daily for 4 to 6 months. In responding patients, maintenance therapy was given at a dose of 3 million units subcutaneously 3 times per week. Responding patients have continued on therapy indefinitely.

ELIGIBILITY:
Age 18-70.

Patients must have morphologically identifiable hairy cells in peripheral blood and bone marrow, or tissue biopsies with at least one of the following: 1) Positive stain for the tartrate-resistant acid phosphatase 2) Electron microscopy compatible with hairy cells.

Patients must be ambulatory with an expected survival greater than 16 weeks and be willing and able to give written informed consent.

Patients must have a disease that is assessable, defined by: 1) Pancytopenia 2) Bone marrow leukemic infiltrate 3) Lymphadenopathy, splenomegaly, or hepatomegaly.

Patients must not require palliative chemotherapy, immunotherapy or hormonal therapy other than the treatment prescribed in this protocol.

Patients must be tested for Hepatitis B surface antigen within one week of entry into this study.

No pregnant or lactating women. No fertile men and women, unless using effective contraception.

No patients with unstable angina. Patients with Class III or IV cardiovascular disease may be entered only after medical clearance by a cardiology consultant.

No patients with severe intercurrent infection or patients having had surgery within the past four weeks unless fully recovered.

No patients with impaired renal function (serum creatinine greater than 1.8).

No patients with impaired hepatic function (total bilirubin greater than 1.4).

No patients with serum calcium greater than 12 mg/dl.

No patients with a performance status less than or equal to 60% on the Karnofsky scale.

No patients who have had any prior (leukocyte or fibroblast) interferon therapy.

No patients unable to carry out the treatment program.

No patients less than 20,000 per cu mm platelets and clinical bleeding disorder; both must be present for patient to be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56
Dates: Start 1997-01; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Knight E Jr, Korant BD. A cell surface alteration in mouse L cells induced by interferon. Biochem Biophys Res Commun. 1977 Jan 24;74(2):707-13. doi: 10.1016/0006-291x(77)90360-6. No abstract available. PMID 836320
- [Background] Lindahl-Magnusson P, Leary P, Gresser I. Interferon and cell division. VI. Inhibitory effect of interferon on the multiplication of mouse embryo and mouse kidney cells in primary cultures. Proc Soc Exp Biol Med. 1971 Dec;138(3):1044-50. doi: 10.3181/00379727-138-36047. No abstract available. PMID 5131604
- [Background] Blomgren H. Steroid sensitivity of the response of human lymphocytes to phytohemagglutinin and pokeweed mitogen: role of phagocytic cells. Scand J Immunol. 1974;3(5):655-64. doi: 10.1111/j.1365-3083.1974.tb01299.x. No abstract available. PMID 4422819